CLINICAL TRIAL: NCT02417207
Title: Entecavir Combined Short-term Intravenous Hepatitis B Immune Globulin (HBIG) to Prevent Hepatitis B Recurrence After Liver Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yang Yang, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (2014)2-127
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis B; Liver Transplantation
Keywords: hepatitis B immune globulin (HBIG); liver transplantation; hepatitis B; entecavir
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Entecavir combined long-term low-dose HBIG group intramuscular (Sham Comparator): HBIG scheme is: the use of intraoperative muscle injection of 800 IU HBIG, postoperative week 1 intramuscular injection HBIG 400 IU 1 times a day, 1 week after intramuscular injection HBIG 400 IU 2 times per week, dosage and time interval according to the HBsAb drops in patients with degree of level adjustment, target drops for 3 months or more after 500 IU/mL, 3 ~ 6 months or 300 IU/mL, after six months of 100 IU/mL or more.
  Interventions: Drug: Entecavir combined long-term low-dose HBIG group intramuscular
- Entecavir combined HBIG group short-term high-dose intravenous (Active Comparator): Preoperative HBV DNA level is less than 1000 IU/ml, intraoperative intravenous drip of 2500 IU HBIG static note type, postoperative 1 and 15 days respectively to give 2500 IU HBIG static note type, a total of three times, then no longer apply. Preoperative HBV DNA level greater than 1000 IU/ml, the use of HBIG solution for: intraoperative intravenous drip of 5000 IU HBIG static note type, postoperative day 1, 15 days and 30 days respectively to give 2000-2500 IU HBIG static note type, a total of four times, since then no longer apply. Preoperative HBV DNA level of the unknown, preoperative immediate detection of DNA, intraoperative intravenous drip of 5000 iu HBIG static note type, choose according to test results after dosing frequency.
  Interventions: Drug: Entecavir combined HBIG group short-term high-dose intravenous

INTERVENTIONS:
Drug: Entecavir combined long-term low-dose HBIG group intramuscular — HBIG scheme is: the use of intraoperative muscle injection of 800 IU HBIG, postoperative week 1 intramuscular injection HBIG 400 IU 1 times a day, 1 week after intramuscular injection HBIG 400 IU 2 times per week, dosage and time interval according to the HBsAb drops in patients with degree of level adjustment, target drops for 3 months or more after 500 IU/mL, 3 ~ 6 months or 300 IU/mL, after six months of 100 IU/mL or more.
  Arms: Entecavir combined long-term low-dose HBIG group intramuscular
Drug: Entecavir combined HBIG group short-term high-dose intravenous — Preoperative HBV DNA level is less than 1000 IU/ml, intraoperative intravenous drip of 2500 IU HBIG static note type, postoperative 1 and 15 days respectively to give 2500 IU HBIG static note type, a total of three times, then no longer apply. Preoperative HBV DNA level greater than 1000 IU/ml, the use of HBIG solution for: intraoperative intravenous drip of 5000 IU HBIG static note type, postoperative day 1, 15 days and 30 days respectively to give 2000-2500 IU HBIG static note type, a total of four times, since then no longer apply. Preoperative HBV DNA level of the unknown, preoperative immediate detection of DNA, intraoperative intravenous drip of 5000 iu HBIG static note type, choose according to test results after dosing frequency.
  Arms: Entecavir combined HBIG group short-term high-dose intravenous

SUMMARY:
The purpose of this study is to observe a new scheme can achieve is the same as the traditional scheme of the effect of preventing hepatitis B recurrence.

DETAILED DESCRIPTION:
At present, the prevention of hepatitis B recurrence after liver transplantation is the most commonly used scheme for nucleoside analogue combined hepatitis B immune globulin (HBIG). HBIG is a condensed to prevent the efficient price of invasion of hepatitis b immunoglobulin, its function is a direct and virus.Also it is to block the virus into liver cells. Lamivudine with HBIG therapy has hepatitis b recurrence rate reduced to below 10%, entecavir combined HBIG hepatitis b recurrence rate is low below 1%. In European and American countries, HBIG the most commonly used method for long-term high-dose intravenous drip, but our country is long-term low-dose intramuscular injection, but all need lifelong medication, for how long after surgery or which patients can disable or not HBIG no consensus. Whether long-term intravenous drip or intramuscular HBIG, are some disadvantages such as high cost, drug side effects, also brought inconvenience to patients. The advent of potent against hepatitis b virus drugs continuously under the background of, in recent years, scholars have already begun to no application or short-term application HBIG discontinuation to prevent hepatitis b recurrence after research, low before transplantation of hepatitis B virus(HBV) DNA replication, such as effective antiviral therapy of hepatitis b recurrence after after transplantation were created the conditions of no HBIG solution. Most studies suggest that transplantation of nucleoside analogues alone for a long time without application or short-term application of HBIG scheme to prevent hepatitis b recurrence is safe, but there are only several transplant center in study abroad, and the Chinese mainland for all application or short-term application of HBIG clinical studies. Entecavir with potent antiviral capacity and high genetic barrier to resistance, low incidence of drug resistance, is currently the prevention and treatment of hepatitis b recurrence after liver transplantation of first-line drugs, entecavir combined long-term muscle injection low-dose HBIG is at present our country is the most commonly used drug for liver transplantation in our center.

This study for entecavir combined after liver transplantation for short-term application type static note HBIG to prevent hepatitis b recurrence of prospective, multicenter, randomized, controlled experimental study, the equivalence. The purpose of this study is to observe a new scheme can achieve is the same as the traditional scheme of the effect of preventing hepatitis B recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. correlation disease hepatitis B viral hepatitis liver transplantation recipients for the first time;
2. older than 18 years old, men and women not limited;
3. preoperative HbsAg positive, regardless of whether preoperative HBV DNA level, regardless of whether preoperative antiviral treatment, regardless of whether associated with primary liver cancer;
4. donor HbsAg negative, other virology negative in liver conditions;
5. to integrate research, good adherence.

Exclusion Criteria:

1. overlap other types of viral hepatitis;
2. the correlation of end-stage liver disease hepatitis b;
3. again to liver transplantation, or joint organ transplantation;
4. allergic to hepatitis b immune globulin;
5. of primary hepatocellular carcinoma with vena cava, portal vein around the trunk or branch, hepatic vein and other large vascular invasion;
6. ABO blood group incompatibility in liver transplantation;
7. moderately severe renal insufficiency, serum creatinine 180 umol/L or higher;
8. there has been a drug resistance of entecavir before liver transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
hepatitis B recurrence after liver transplantation | 2years

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yang, MD, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Wang Guoying, Guangzhou, Guangdong, China